CLINICAL TRIAL: NCT06423924
Title: Risk Factors, Cancer Types and Prognostic Significance of Second Primary Cancer Based on the Early-onset and Late-onset Colorectal Cancer
Brief Title: Second Primary Cancer and Early-onset Colorectal Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: LI XIN-XIANG (Other)
Responsible Party: Sponsor-Investigator, LI XIN-XIANG, professor, Fudan University
Organization: Fudan University (Other)
Other Study IDs: CRCSPM
Record Dates: First submitted 2024-05-11; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Colorectal Cancer; Second Primary Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms, Second Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- <50 years
  Interventions: Other: no intervention
- 50-69 years
  Interventions: Other: no intervention
- ≥70 years
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The objective of this study was to analyze the pathological factors influencing the occurrence and prognosis of SPC in CRC patients of varying ages and compare the differences in the patterns of SPC occurrence and prognosis among patients of different age groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing radical surgery for colorectal cancer at Fudan University Shanghai Cancer Center between January 2008 and December 2018.
* Stage Ⅰ-Ⅳ colorectal cancer confirmed by clear pathological information

Exclusion Criteria:

* Previous history of other cancers before surgery
* Patients under 18 years old or over 80 years old

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients retrieved from the database of Fudan University Shanghai Cancer Center. These patients were diagnosed with CRC primary tumors between January 2008 and December 2018.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-05-11 (Estimated); Primary Completion 2024-05-20 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | The duration from the date of surgery to death for any reason or the last recorded follow-up, whichever comes first. Up to 100 months
  The duration from the date of surgery to death for any reason or the last recorded follow-up, whichever comes first.
  Up to 100 months

IPD SHARING:
Plan to Share IPD: No